CLINICAL TRIAL: NCT00612846
Title: A Randomised Clinical Trial to Compare Endoscopic Sphincterotomy and Subsequent Laparoscopic Cholecystectomy With Primary Laparoscopic Bile Duct Exploration During Cholecystectomy in Higher Risk Patients With Choledocholithiasis
Brief Title: Study Investigating the Best Method of Treatment of Bile Duct Stones in Higher Risk Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated early due to slow recruitment
Sponsor: North Bristol NHS Trust (Other)
Responsible Party: Michael H Thompson, North Bristol NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112/99
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Choledocholithiasis; Higher Risk Patients
Keywords: Common Bile Duct Calculi; Choledocholithiasis; Endoscopic sphincterotomy; Cholecystectomy, laparoscopic; Laparoscopic bile duct exploration
MeSH Terms: conditions — Choledocholithiasis; Gallstones | interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Procedure: Endoscopic sphincterotomy and subsequent laparoscopic cholecystectomy
- B (Experimental)
  Interventions: Procedure: Laparoscopic bile duct exploration during cholecystectomy

INTERVENTIONS:
Procedure: Endoscopic sphincterotomy and subsequent laparoscopic cholecystectomy — Endoscopic sphincterotomy and subsequent laparoscopic cholecystectomy
  Arms: A
Procedure: Laparoscopic bile duct exploration during cholecystectomy — Laparoscopic bile duct exploration during cholecystectomy
  Arms: B

SUMMARY:
The aim of the trial is to compare two operations which are used to treat bile duct stones. The hypothesis of the study is that there is no difference between endoscopic sphincterotomy followed by laparoscopic cholecystectomy or laparoscopic bile duct exploration during laparoscopic cholecystectomy in the treatment of bile duct stones in higher risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Gallbladder stones
* At least strong evidence of bile duct stones (abnormal LFTs and dilated bile duct)
* Higher risk (>70yrs, >60yrs with co-morbidity, >50 with BMI>40)

Exclusion Criteria:

* Not fit for general anaesthesia
* Cholangitis requiring emergency ERCP
* Previous upper GI surgery making ERCP impossible

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2000-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Bile duct clearance | Peri-operative

SECONDARY OUTCOMES:
Morbidity and mortality | 30 day or directly relating to intervention
Post-operative stay | Post-operative stay
Procedures per patient | Interventions required to acheive duct clearance
Conversion to open surgery | Peri-operative

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Thompson, MD, FRCS, Study Director — North Bristol NHS Trust